CLINICAL TRIAL: NCT06849843
Title: A Multicenter, Randomized, Controlled Clinical Study of 3mg Once Every Two Weeks Administration of Efsubaglutide Alfa Injection in Type 2 Diabetes Patients With Poor Glycemic Control After Diet and Exercise Intervention.
Brief Title: A Study of 3mg Once Every Two Weeks Administration of Efsubaglutide Alfa Injection in Type 2 Diabetes Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YN011-201
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3mg of Efsubaglutide Alfa QoW (Experimental)
  Interventions: Drug: Efsubaglutide Alfa Injection
- 1mg of Efsubaglutide Alfa QW (Active Comparator)
  Interventions: Drug: Efsubaglutide Alfa Injection

INTERVENTIONS:
Drug: Efsubaglutide Alfa Injection — Efsubaglutide Alfa 3mg/0.5ml
  Arms: 3mg of Efsubaglutide Alfa QoW
Drug: Efsubaglutide Alfa Injection — Efsubaglutide Alfa 1mg/0.5ml
  Arms: 1mg of Efsubaglutide Alfa QW

SUMMARY:
This is a study to evaluate the impact and efficacy of Efsubaglutide Alfa injection 3mg QoW on the treatment of type 2 diabetes patients with poor glycemic control after dietary and exercise intervention.

Primary objective:

To evaluate the effect and role of continuous treatment with 3mg of Efsubaglutide Alfa QoW and 1mg of Efsubaglutide Alfa QW for 12 weeks on HbA1c in T2DM patients with poor glycemic control after dietary and exercise intervention.

Secondary objectives:

1. To evaluate the effect of continuous treatment with 3mg of Efsubaglutide Alfa QoW for 12 weeks on glucose variability (change in time in range (TIR) relative to baseline) in T2DM patients with poor glycemic control after dietary and exercise intervention.
2. To evaluate the effect of continuous treatment with 3mg of Efsubaglutide Alfa QoW for 12 weeks on drug exposure (relative to 1mg QW) in T2DM patients with poor glycemic control after dietary and exercise intervention.
3. To evaluate the effect of continuous treatment with 3mg of Efsubaglutide Alfa QoW for 12 weeks on fasting plasma glucose (FPG) in T2DM patients with poor glycemic control after dietary and exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 18 to 75;
2. Type 2 diabetes diagonsed at least 8 weeks and has not received any glucose-lowering medication within 8 weeks prior to screening;
3. During screening, HbA1c: 7.0% ≤ HbA1c ≤ 11.0%;
4. Before randomization : 7.0% ≤ HbA1c ≤ 11.0%;
5. During screening and before randomization: FPG< 13.9 mmol/L
6. 24 kg/m2 ≤ BMI ≤ 40 kg/m2;
7. Without birth plan and voluntarily take effective contraceptive measures;
8. Fully understood the study, voluntarily entered the study and signed the informed consent.

Exclusion Criteria:

1. Diabetes other than Type 2;
2. Any DPP-4 inhibitors and / or GLP-1 analogues were used within 3 months before screening;
3. Continuous use of insulin for more than 14 days in the previous year;
4. C-Peptide <0.3 nmol/L;
5. Diabetic ketoacidosis, diabetic lactic acidosis or hyperosmolar non ketonic diabetic coma occurred within 6 months before screening;
6. Unstable proliferative retinopathy or macular lesion, severe diabetic neuropathy, intermittent claudication or diabetic foot occurred within 6 months before screening;
7. Severe hypoglycemia occurred within 6 months before screening
8. Severe trauma infection or operation within one month before screening;
9. Blood donation or massive blood loss or transfusion within 3 months ;
10. Suspected active infection ;
11. Growth hormone therapy was performed within 6 months before screening;
12. Patients having received corticosteroid continuous ≥ 7 days through within 2 months ;
13. Use any drugs or surgery with weight control effect within 2 months;
14. weight change of more than 5% within 3 months;
15. mean systolic pressure (SBP) ≥ 160mmhg and / or DBP ≥ 90 mmHg at screening, or new/changed antihypertensive drugs or adjusted dosage of antihypertensive drugs within 4 weeks before screening or before induction period
16. with a history of severe cardiovascular disease, high risk of stroke/stroke within 6 months before screening;
17. with a history of acute or chronic pancreatitis, symptomatic gallbladder , pancreatic injury and other risk factors for pancreatitis, or with blood amylase and/or blood lipase ≥1.5 times the upper limit of normal (ULN) at the time of screening or before randomization;
18. Calcitonin level ≥50 ng/L (pg/mL) during screening;
19. with a history of medullary thyroid cancer, multiple endocrine neoplasm (Men) 2A or 2B syndrome, or related family history;
20. with clinically significant abnormal gastric emptying , severe chronic gastrointestinal diseases , long-term use of drugs that have a direct impact on gastrointestinal peristalsis , or having undergone gastrointestinal surgery within 6 months before screening, are not suitable to participate in this clinical study according to the evaluation of the researchers;
21. suffering from hematological diseases or any disease causing hemolysis or erythrocyte instability ;
22. Uncontrolled hyperthyroidism or hypothyroidism;
23. with hemoglobinopathy that may affect the determination of HbA1c levels;
24. HBsAg, HCV-Ab, HIV-Ab, TPAb or COVID-19 nucleic acid tested positive;
25. serious mental illness;
26. drinking more than 14 standard units weekly within 6 months before screening ;
27. a history of organ transplantation or other acquired or congenital immune system diseases;
28. allergic to the active ingredients (GLP-1 and GLP-1 analogues) of the study drug;
29. clear contraindications for the use of metformin;
30. Any of the following conditions: the pacemaker was installed when screened; no pacemaker was installed, but 12 lead ECG showed degree II or III atrioventricular block, long QT syndrome or QTc interval ≥ 450ms (fridericia formula was used to calculate QTCF); Patients with New York Heart Function Classification III or IV; Or other abnormal cardiac function with clinical significance that is not suitable for clinical research judged by researchers;
31. acute or chronic viral hepatitis, or whose laboratory examination indexes meet one of the following criteria at the time of screening or before randomization : alanine aminotransferase (ALT) level ≥ 2.5 fold ULN, aspartate aminotransferase (AST) ≥ 2.5 fold ULN, fasting triglyceride (TG) > 5.7 mmol/L or 500 mg/dl; the glomerular filtration rate (EGFR) < 60 ml/min/1.73 m2 was calculated by CKD-EPI (epi - (SCR)) formula;
32. participated in clinical trials of other drugs or devices within 3 months before screening;
33. Medication compliance in the lead-in period was ≤ 50% ;
34. Any other situation that researchers think may affect the patients' informed consent or compliance with the trial protocol, or the patients' participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  The change in mean HbA1c concentrations (%)from baseline with Efsubaglutide Alfa 3mg QoW versus Efsubaglutide Alfa 1mg QW

SECONDARY OUTCOMES:
TIR | 12 weeks
  Changes in the percentage of time in range (TIR) relative to baseline
HbA1c<7.0% and <6.5% | 12 weeks
  The proportion of participants who achieved HbA1c target (HbA1c<7.0% and <6.5% Patient percentage)
fasting lipid profiles | 12 weeks
  Changes in fasting lipid(TC/TG/HDL-C/LDL-C) profiles relative to baseline(mmol/L)
weight | 12 weeks
  Weight change from baseline(kg)
waist circumference | 12 weeks
  Absolute changes in waist circumference(cm) from baseline
hip circumference | 12 weeks
  Absolute changes in hip circumference(cm) from baseline
waist-to-hip ratio (WHR) | 12 weeks
  Absolute changes in waist-to-hip ratio (WHR) from baseline
salvage treatment | 12 weeks
  Percentage of subjects receiving salvage treatment(%)
body fat composition | 12 weeks
  Changes in body fat composition from baseline
FPG | 12 weeks
  Changes in FPG (mmol/L) relative to baseline

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Nanjing First Hospital, Nanjing, Jiangsu
  - CangZhou Hospital of Integrated TCM and Western Medicine in Hebei Province, Cangzhou
  - Huzhou Central Hospital, Huzhou
  - Jiangsu Province Offical Hospital, Nanjing
  - Ningbo First Hospital, Ningbo
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou Central Hospital, Wenzhou
  - Zibo Municipal Hospital, Zibo